CLINICAL TRIAL: NCT06780085
Title: KEYMAKER-U01 Substudy 01H: A Phase 2, Randomized, Umbrella Study With Rolling Arms of Investigational Agents in Participants With Previously Treated Stage IV Nonsquamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Investigational Agents in Participants With Previously Treated Stage IV Nonsquamous Non-small Cell Lung Cancer (NSCLC) (MK-3475-01H/KEYMAKER-U01)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-01H; 2024-518761-10-00 (Registry Identifier: EU CT); MK-3475-01H (Other: MSD); U1111-1314-1785 (Registry Identifier: UTN); KEYMAKER-U01 (Other: MSD)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Unblinded open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Raludotatug Deruxtecan (Experimental): Participants receive raludotatug deruxtecan (R-DXd) 5.6 mg/kg via intravenous (IV) Infusion every 3 weeks (q3w) until disease progression or discontinuation criterion is met.
  Interventions: Biological: Raludotatug Deruxtecan
- Ifinatamab Deruxtecan (Experimental): Participants receive ifinatamab deruxtecan (I-DXd) 12 mg/kg via IV infusion q3w until disease progression or discontinuation criterion is met.
  Interventions: Biological: Ifinatamab Deruxtecan
- Docetetaxel (Active Comparator): Participants receive docetaxel 75mg/m2 via IV infusion q3w until disease progression or discontinuation criterion is met.
  Interventions: Drug: Docetetaxel

INTERVENTIONS:
Biological: Raludotatug Deruxtecan — IV Infusion
  Other Names: R-DXd; MK-5909; DS-6000a
  Arms: Raludotatug Deruxtecan
Biological: Ifinatamab Deruxtecan — IV Infusion
  Other Names: I-DXd; MK-2400; DS-7300a
  Arms: Ifinatamab Deruxtecan
Drug: Docetetaxel — IV Infusion
  Arms: Docetetaxel

SUMMARY:
Researchers are looking for new ways to treat metastatic nonsquamous non-small cell lung cancer (NSCLC) that has been treated before. Metastatic means the cancer has spread to other parts of the body. Nonsquamous means the cancer did not start in squamous cells, which are flat cells that line the inside of the lungs.

Standard treatment (usual treatment) for NSCLC is surgery, then immunotherapy with or without chemotherapy after surgery. Immunotherapy is a treatment that helps the immune system fight cancer. Chemotherapy is a medicine that works to destroy cancer cells or stop them from growing.

However, standard treatment may not work or may stop working for some people. Researchers want to know if 2 antibody drug conjugates (ADCs) can help treat metastatic nonsquamous NSCLC that did not respond (get smaller or go away) to treatment. An ADC attaches to specific targets on cancers cells and delivers treatment to destroy those cells.

Researchers will compare 2 different ADCs (the study treatments) to chemotherapy in this study. The goals of this study are to learn:

* About the safety of the study treatments and if people tolerate them
* How many people have the cancer respond to the study treatments

DETAILED DESCRIPTION:
The master screening protocol is MK-3475-U01 (KEYMAKER-U01) - NCT04165798

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Histologically or cytologically confirmed diagnosis of Stage IV nonsquamous non-small cell lung cancer (NSCLC)
* Documented disease progression per RECIST 1.1 after receiving an anti-programmed cell death 1 protein (PD-1)/programmed cell death ligand 1 (PD-L1) treatment and platinum-based chemotherapy
* Confirmation per local test report that epidermal growth factor receptor negative (EGFR-), anaplastic lymphoma kinase negative (ALK-), or c ros oncogene 1 negative (ROS1-) directed therapy is not indicated as primary therapy
* Measurable disease per RECIST 1.1 as assessed by investigator and verified by BICR
* Life expectancy of at least 3 months
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before randomization
* Is an individual of any sex/gender who is at least 18 years of age at the time of providing the informed consent
* Has adequate organ function
* If capable of producing sperm refrains from donating sperm plus either abstains from penile-vaginal intercourse or uses a penile/external condom, with contraceptive use consistent with local regulations
* Participant/participants of childbearing potential (POCBP) is not pregnant and has a negative highly sensitive pregnancy test; and is not breastfeeding and uses a highly effective contraceptive method
* Archival tumor tissue sample of a tumor lesion not previously irradiated has been provided
* Has provided tissue prior to treatment randomization from a newly obtained formalin-fixed sample from a new biopsy
* Human Immunodeficiency Virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Received radiation therapy to the lung
* Has uncontrolled or significant cardiovascular disorder prior to randomization
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Participants who have adverse events (AEs) (other than alopecia) due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline
* Has known severe hypersensitivity (≥Grade 3) to study intervention and/or any of its excipients
* Has evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection (including HIV infection)
* Has clinically significant corneal disease
* Has received prior radiotherapy within 2 weeks of start of study intervention, or radiation related toxicities, requiring corticosteroids
* Has inadequate washout period prior to randomization
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has evidence of any leptomeningeal disease
* Has history of (noninfectious) pneumonitis/ interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD, and/or suspected ILD/pneumonitis
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has active infection requiring systemic therapy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease
* Has known history of, or active, neurologic paraneoplastic syndrome
* Has history of allogeneic tissue/solid organ transplant
* Have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2032-03-12 (Estimated); Study Completion 2032-03-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 81 months
  ORR is defined as the percentage of participants with Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Percentage of Participants with at Least One Adverse Event (AE) | Up to approximately 81 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The percentage of participants who experience an AE will be reported.
Percentage of Participants Who Discontinued Medication Due to an AE | Up to approximately 24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The percentage of participants who discontinue study intervention due to an AE will be reported.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 81 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-free Survival (PFS) | Up to approximately 81 months
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 81 months
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- United States (2):
  - University of Kentucky Chandler Medical Center ( Site 0019), Lexington, Kentucky
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
- Chile (3):
  - Centro de Estudios Clínicos SAGA ( Site 0161), Santiago, Region M. de Santiago
  - FALP ( Site 0160), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0162), Santiago, Region M. de Santiago
- Germany (2):
  - Universitaetsklinik Tuebingen ( Site 0192), Tübingen, Baden-Wurttemberg
  - Charite-Universitaetsmedizin Berlin ( Site 0191), Berlin
- Greece (2):
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 0204), Athens, Attica
  - European Interbalkan Medical Center ( Site 0205), Thessaloniki
- Hungary (3):
  - Bacs-Kiskun Varmegyei Oktatokorhaz ( Site 0063), Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz ( Site 0062), Győr, Győr-Moson-Sopron
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Gyula Korhaz-Rendelointezet ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
- Israel (6):
  - Rambam Health Care Campus ( Site 0076), Haifa
  - Shaare Zedek Medical Center ( Site 0075), Jerusalem
  - Meir Medical Center ( Site 0071), Kfar Saba
  - Rabin Medical Center ( Site 0074), Petah Tikva
  - Sheba Medical Center ( Site 0070), Ramat Gan
  - Sourasky Medical Center ( Site 0077), Tel Aviv
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0175), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi ( Site 0173), Florence
  - Ospedale San Raffaele. ( Site 0171), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 0174), Roma
- Poland (4):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii ( Site 0153), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie ( Site 0152), Koszalin, West Pomeranian Voivodeship
- Hospital Universitario Quiron Madrid ( Site 0091), Madrid, Spain
- Turkey (Türkiye) (2):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 0140), Ankara
  - I. U. Cerrahpasa Tip Fakultesi ( Site 0144), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com